CLINICAL TRIAL: NCT04285879
Title: A Determination of Efficacy and Therapeutic Benefits of Blood Flow Restriction Training in an Adolescent Population
Brief Title: Blood Flow Restriction Training (BFR) in an Adolescent Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Principal Investigator, Adam Weaver, Physical Therapist, Connecticut Children's Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-168
Record Dates: First submitted 2020-02-20; First posted 2020-02-26 (Actual); Results first posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Blood Flow Restriction; ACL Tear; ACL Injury
Keywords: physical therapy; rehabilitation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: The investigators will compare the use of exercises augmented with BFR with quantitative measurements of strength and patient reported outcomes. A total of 20 youth and adolescent patients undergoing a surgical procedure for ACL reconstruction at Connecticut Children's Elite Sports Medicine and completing physical therapy at Connecticut Children's Sports Physical Therapy will be recruited for this study. A review of data from 20 previous patients, matched for age, sex, BMI and surgical procedure that completed physical therapy at Connecticut Children's Sports Physical Therapy will be used as a comparison.
  As part of this pilot study, the investigators will additionally collect prospective controls. This population will be patients not participating in physical therapy at Connecticut Children's but underwent ACL reconstruction by Elite Sports Medicine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- BFR Exercise Group (Experimental): In addition to the standard ACL protocol, patients in this study will utilize the Owen Recovery Science exercise protocol for BFR [18]. The following guidelines will be followed concerning exercise progression, occlusion pressure and difficulties with volume achievement.
  A total of 20 youth and adolescent patients undergoing a surgical procedure for ACL reconstruction at Connecticut Children's Elite Sports Medicine and completing physical therapy at Connecticut Children's Sports Physical Therapy will be recruited for this study.
  Interventions: Device: Blood Flow Restriction using Delfi Personalized Tourniquet System
- Non-BFR exercise group (No Intervention): As part of this pilot study, the investigators will additionally collect prospective controls. This population will be patients not participating in physical therapy at Connecticut Children's but underwent ACL reconstruction by Elite Sports Medicine

INTERVENTIONS:
Device: Blood Flow Restriction using Delfi Personalized Tourniquet System — The Delfi Tourniquet System is designed to be used in conjunction with exercise. The system automatically determines the degree of occlusion and allows for safe regulation of pressure. Patients will then complete exercises with the use of this device following the Owens Recovery Science Protocol
  Other Names: FDA Establishment Registration Number 9681444. Device Listing Number E127474. Classification Number 878.5910. Product Code KCY. 510(k) Exempt. MID: XCDELMED1099VAN
  Arms: BFR Exercise Group

SUMMARY:
While there are a number studies that have reported on the use of BFR in the adult population, there is limited information about the use of BFR in the adolescent population. This study aims to evaluate the use of BFR training in conjunction with traditional ACL (anterior cruciate ligament) reconstruction rehabilitation in adolescents.

The purpose of this study is to evaluate the addition of BFR-based exercise to traditional methods of physical therapy. Does the use of BFR-based exercise improve strength, hypertrophy, functional and patient reported outcomes after ACL Reconstruction in the adolescent population?

DETAILED DESCRIPTION:
The planned pilot study is a prospective case control study utilizing retrospective controls. The investigators will compare the use of exercises augmented with BFR with quantitative measurements of strength and patient reported outcomes. A total of 20 youth and adolescent patients undergoing a surgical procedure for ACL reconstruction at Connecticut Children's Elite Sports Medicine and completing physical therapy at Connecticut Children's Sports Physical Therapy will be recruited for this study. A review of data from 20 previous patients, matched for age, sex, BMI and surgical procedure that completed physical therapy at Connecticut Children's Sports Physical Therapy will be used as a comparison.

As part of this pilot study, the investigators will additionally collect prospective controls. This population will be patients not participating in physical therapy at Connecticut Children's, but underwent ACL reconstruction by Elite Sports Medicine. The investigators are unsure of the ability for us to collect prospective controls in a timely manner, hence the investigators will use the above described retrospective cohort as controls if the prospective controls prove difficult to recruit.

Identification and Recruitment:

All potential patients undergoing ACL reconstruction at Elite Sports Medicine will be approached for participation for this study. Eligible patients will be identified at their initial pre-operative appointment with the Sports Medicine Physician, Athletic Trainer, and Sports Physical Therapy Physical Therapist. Subject selection will be completed by those patients meeting the above outlined inclusion and exclusion criteria. At this time, the study purpose and protocol will be explained and a brief summary of the study will be provided.

Consent: Consent will take place at the pre-operative visit. The patient/parent will be given a detailed description of the purpose and methodology for this study. The participants will have the opportunity to read the consent forms and ask any questions they may have about the research. If the patients agree to participate, they will be asked to sign the consent form and a copy will be provided.

Retention: Eligible patients will be required to be seen for a minimum of 90% of patient visits to be included in this study.

In addition to the standard ACL protocol, patients in this study will utilize the Owen Recovery Science exercise protocol for BFR [18]. The following guidelines will be followed concerning exercise progression, occlusion pressure and difficulties with volume achievement. To determine the appropriate resistance for each exercise, the patient's 1 repetition maximum (1RM) will be attained using a repetition test [19]. This test will use a previously validated algorithm to determine the 1RM based on the weight used to perform a 7-10 repetition test [20]. Patient will perform the exercise with a weight they can comfortably lift for several repetitions. Based on the weight or resistance used, and the patient's perceived exertion a 1RM will be estimated using the modified OMNI-RES (OMNI perceived exertion scale for resistance). The starting load for each exercise will be 20-30% of their 1RM , or bodyweight resistance will be used when loading is not feasible.

Proposed Protocol Phase 1- Weeks 1 to 2

* Quad Set: 10 second on, 10 second rest at 100% occlusion x10'

  o progress to isometrics at the edge of the table 60 degrees as clinically appropriate
* Side Lying Hip Abduction, 30/15/15/15, at 80% occlusion
* Hip Extension from prone 30/15/15/15, at 80% occlusion
* Re-check load at the start of each Phase, to determine 1 RM (7-10 RM (repetition maximum) test on leg press)
* Total BFR time approximately 24 minutes per session, with 2 sessions per week

Phase 2- Weeks 3 to 4

* Replace Quad Set with Long Arc Quad (90-30deg), 30/15/15/15 at 80% occlusion
* Replace Hip Extension with Leg Press (shuttle), 30/15/15/15 at 80% occlusion
* Hip Abduction, 30/15/15/15 at 80% occlusion
* Total BFR time approximately 24 minutes per session with 2 sessions per week

Phase 3- Weeks 5 to 6

* Long Arc Quad (90-30deg), 30/15/15/15 at 80% occlusion
* Leg Press (shuttle), 30/15/15/15 at 80% occlusion
* Replace Hip Abduction with Bilateral Hip Bridge, 30/15/15/15 at 80% occlusion
* Total BFR time approximately 24 minutes per session, with 2 sessions per week

Phase 4- Weeks 7 to 8

* Leg Press (shuttle), 30/15/15/15 at 80% occlusion
* Replace Long Arc Quad with Step Up 30/15/15/15 at 80% occlusion
* Bilateral Hip Bridge, 30/15/15/15 at 80% occlusion
* Total BFR time approximately 24 minutes per session, with 2 sessions per week

Phase 5- Weeks 9 to 12

* Replace Bilateral Hip Bridge with Medial Step Down, 30/15/15/15 at 80% occlusion
* Replace Step up with Split Squat, 30/15/15/15 at 80% occlusion
* Leg Press (shuttle), 30/15/15/15 at 80% occlusion
* Total BFR time approximately 24 minutes per session, with 2 sessions per week

Phase 6- Weeks 11 to 12

* Progressively load exercises from phase 5
* Total BFR time approximately 24 minutes per session, with 2 sessions per week

ELIGIBILITY:
Inclusion Criteria:

* Patients between the age of 12 and 18 years at the time of surgery.
* Post-primary ACL reconstruction
* Orthopaedic surgical intervention (including all additional procedures at the knee) completed by one of the Elite Sports Medicine physicians.
* Patient completed postoperative rehabilitation following standard protocols
* No contraindications to performing BFR, as outlined in the Owens Recovery[18] Science 2018 Personal Blood Flow Restriction manual.

Exclusion Criteria:

* Patients older than 18 and younger than 12 at the time of surgery
* Any additional diagnoses or deformity not related to knee injury that could affect knee strength
* Additional lower extremity injury at time of knee injury (e.g., ankle injury) requiring treatment
* Previous surgical intervention on the knee (ipsilateral and contralateral)
* Patients with weight bearing restrictions for greater than two weeks after surgery due to concomitant pathology such as meniscal root/radial repair, chondral pathology, or multi-ligament pathology. . Generic exclusion: "Subjects not meeting all inclusion criteria."

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Weaver, PT, DPT, Principal Investigator — Physical Therapist
Locations (1):
- Connecticut Children's Sports Physical Therapy, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- BFR Exercise Group: In addition to the standard ACL protocol, patients in this study will utilize the Owen Recovery Science exercise protocol for BFR [18]. The following guidelines will be followed concerning exercise progression, occlusion pressure and difficulties with volume achievement.
  A total of 20 youth and adolescent patients undergoing a surgical procedure for ACL reconstruction at Connecticut Children's Elite Sports Medicine and completing physical therapy at Connecticut Children's Sports Physical Therapy will be recruited for this study.
  Blood Flow Restriction using Delfi Personalized Tourniquet System: The Delfi Tourniquet System is designed to be used in conjunction with exercise. The system automatically determines the degree of occlusion and allows for safe regulation of pressure. Patients will then complete exercises with the use of this device following the Owens Recovery Science Protocol
- Non-BFR Exercise Group: As part of this pilot study, the investigators will additionally collect prospective controls. This population will be patients not participating in physical therapy at Connecticut Children's but underwent ACL reconstruction by Elite Sports Medicine. Per our IRB protocol, should we be unable to obtain prospective controls a review of prior patients from previous patients matched for age, sex and Surgical procedure to provide a retrospective cohort.
Period: Overall Study
Arm/Group | BFR Exercise Group | Non-BFR Exercise Group
Started | 33 | 14
Completed | 16 | 6
Not Completed | 17 | 8
Not completed — Lost to Follow-up | 1 | 8
Not completed — medical/surgical exclusion | 16 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BFR Exercise Group | Non-BFR Exercise Group | Total
Number analyzed (Participants) | 33 | 14 | 47
Age, Continuous [Mean (Full Range); unit: years] | 15.46 [12.45 to 18.42] | 15.33 [12.45 to 17.50] | 15.43 [12.45 to 18.42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 9 | 29
  Male | 13 | 5 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Full Range); unit: inches] | 65.64 [61 to 74] | 65.66 [63 to 74] | 65.65 [61 to 74]
weight [Mean (Full Range); unit: lbs] | 146 [96 to 228] | 165 [110 to 291] | 151 [96 to 291]

OUTCOME MEASURES:

1. Primary Outcome: Isometric Quad Strength Peak Torque
Description: Isometric strength testing to measure peak torque quadriceps strength (unit: nm/kg) as reported by isokinetic dynamometer on involved and uninvolved limb.
Time Frame: 3 month and return to sport post-operative strength (6-8 months post-op)
Population: We enrolled 47 patients in our study. Due to exclusion criteria, patients lost to follow up and COVID-19 pandemic we were unable to fully analyze all consented patients in both groups.
Measure: Mean (Standard Deviation); unit: Nm/kg
Groups:
- Non-BFR Exercise Group: As part of this pilot study, the investigators will additionally collect prospective controls. This population will be patients not participating in physical therapy at Connecticut Children's but underwent ACL reconstruction by Elite Sports Medicine.
  due to limitations in our prospective control, we use an aged match retrospective cohort of 16 patients for analysis.
Arm/Group | BFR Exercise Group | Non-BFR Exercise Group
Number analyzed (Participants) | 33 | 14
Nm/kg
  3 month isometric: number analyzed (Participants) | 16 | 11
  3 month isometric | 1.83 (.35) | 1.31 (0.63)
  return to sport isometric (between approximately 6-8 months post-op): number analyzed (Participants) | 33 | 5
  return to sport isometric (between approximately 6-8 months post-op) | 2.45 (0.64) | 2.1 (0.6)

2. Primary Outcome: Isometric Quad Strength Limb Symmetry Index
Description: Quadriceps limb symmetry index is calculated by taking the values from outcome 1. [ ( peak torque quadriceps involved limb (nm-kg)/ peak torque quadriceps uninvolved limb (nm-kg))*100] as reported by isokinetic dynamometer. This value is expressed as a percentage. 100% would equal perfect symmetry. Should involve limb demonstrate greater strength then uninvolved limb symmetry scores would be greater then 100%
Time Frame: 3 month and return to sport isometric quad strength limb symmetry
Population: We enrolled 47 patients in our study. Due to exclusion criteria, patients lost to follow up and COVID-19 pandemic we were unable to use all patients that were consented for analysis.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | BFR Exercise Group | Non-BFR Exercise Group
Number analyzed (Participants) | 33 | 14
percent
  3 month post-op: number analyzed (Participants) | 16 | 11
  3 month post-op | 68.02 (13.94) | 60.72 (17.54)
  Return to sport (@ 6-8 months post-op): number analyzed (Participants) | 16 | 5
  Return to sport (@ 6-8 months post-op) | 89.53 (27.74) | 80.97 (10.69)

3. Primary Outcome: Isometric Hamstring Strength Peak Torque
Description: Isometric strength testing to measure peak torque hamstring strength (unit:nm/kg) as reported by isokinetic dynamometer on involved and uninvolved limb.
Time Frame: at 3 months post-op and return to sport (between approximately 6-8 months post-op)
Population: We enrolled 47 patients in our study. Due to exclusion criteria, patients lost to follow up and COVID-19 pandemic we were unable to use all data for consented subjects in both groups.
Measure: Mean (Standard Deviation); unit: nm/kg
Arm/Group | BFR Exercise Group | Non-BFR Exercise Group
Number analyzed (Participants) | 33 | 14
nm/kg
  3 months post-op: number analyzed (Participants) | 33 | 11
  3 months post-op | 1.20 (0.51) | 1.61 (0.36)
  return to sport (between approximately 6-8 months post-op): number analyzed (Participants) | 33 | 5
  return to sport (between approximately 6-8 months post-op) | 1.53 (0.30) | 1.3 (0.41)

4. Primary Outcome: Isometric Hamstring Strength Limb Symmetry Index
Description: Hamstring limb symmetry index is calculated by taking the values from outcome 3 [ ( peak torque hamstring involved limb (nm-kg) / peak torque hamstring uninvolved limb (nm-kg))*100] as reported by isokinetic dynamometer. This value is expressed as a percentage.100% would equal symmetry. For patients that demonstrate a stronger involved limb then uninvolved limb symmetry will be reported as greater then 100%
Time Frame: 3 months post op and return to sport (between approximately 6-8 months post-op)
Population: We enrolled 47 patients in our study. Due to exclusion criteria, patients lost to follow up and COVID-19 pandemic we were unable to use data for all consented patients for both groups.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | BFR Exercise Group | Non-BFR Exercise Group
Number analyzed (Participants) | 33 | 14
percent
  3 months post-op: number analyzed (Participants) | 33 | 11
  3 months post-op | 108.32 (21.41) | 80.3 (14.71)
  return to sport (between approximately 6-8 months post-op): number analyzed (Participants) | 33 | 5
  return to sport (between approximately 6-8 months post-op) | 96.74 (11.68) | 85.61 (16.21)

5. Secondary Outcome: Pedi-IKDC (International Knee Documentation Committee)
Description: Patient Reported Outcome Measure- Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
Time Frame: at 3 months post-op and return to sport (between approximately 6-8 months post-op)
Population: We enrolled 47 patients in our study. Due to exclusion criteria, patients lost to follow up and COVID-19 pandemic we were unable to use all data for all consented patients in both groups
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BFR Exercise Group | Non-BFR Exercise Group
Number analyzed (Participants) | 33 | 14
units on a scale
  3 months: number analyzed (Participants) | 33 | 11
  3 months | 68.91 (9.68) | 71.82 (16.78)
  return to sport (between approximately 6-8 months post-op): number analyzed (Participants) | 33 | 5
  return to sport (between approximately 6-8 months post-op) | 89.42 (7.94) | 80.90 (8.04)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the study time period when patients were completing BFR training during their physical therapy session for 12 weeks.
Description: monitoring for the following side effects: subcutaneous hemorrhage (SubQ), deep vein thrombosis (DVT), fainting, dizziness, lower extremity paresthesia, and itching
Arm/Group | BFR Exercise Group | Non-BFR Exercise Group
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/14
Other Adverse Events (participants affected / at risk) | 0/33 | 0/14

LIMITATIONS AND CAVEATS:
Covid-19 pandemic Lost to follow up, surgical exclusion led to small number of controls.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/79/NCT04285879/Prot_SAP_001.pdf